CLINICAL TRIAL: NCT07093138
Title: Evaluation of Efficacy and Safety of Topical Cannabidiol (Canvert-M Produced by Alasht Pharmed co. Iran) in the Treatment of Migraine Attacks
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alasht Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CANM.ALA.MT.IV.O3
Record Dates: First submitted 2025-07-20; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Migraine Disorders
Keywords: Cannabidiol; Migraine disorders; Mentha piperita; Lavandula; Eucalyptus; Ocimum basilicum; Rosmarinus; Gaultheria; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canvert-M (Produced by Alasht Pharmed co. Iran) (Experimental): Canvert-M is a topical roll-on formulation that contains cannabidiol, peppermint, lavender, rosemary, eucalyptus, wintergreen, basil oil, etc. At the onset of a migraine attack, an adequate amount of Canvert-M roll-on should be applied to the areas of the forehead, temporal, behind the ears, and the base of the neck.
  Interventions: Combination Product: Canvert-M (Produced by Alasht Pharmed co. Iran)

INTERVENTIONS:
Combination Product: Canvert-M (Produced by Alasht Pharmed co. Iran) — Canvert-M is a topical roll-on formulation that contains cannabidiol, peppermint, lavender, rosemary, eucalyptus, wintergreen, basil oil, etc. At the onset of a migraine attack, an adequate amount of Canvert-M roll-on should be applied to the areas of the forehead, temporal, behind the ears, and the base of the neck. If the patient's headache persists after 30 minutes, a second dose can be used.

SUMMARY:
Canvert-M (manufactured by Alasht Pharmed Co. Iran) is a topical roll-on formulation that contains cannabidiol, peppermint, lavender, rosemary, eucalyptus, wintergreen, basil oil, etc. This phase IV, single-arm, open-label clinical trial evaluated the efficacy and safety of Canvert-M in males and females aged 18 to 55 years diagnosed with migraine according to the International Classification of Headache Disorders, 3rd edition (ICHD-3), for the treatment of migraine attacks.

The primary objective was to assess the reduction in headache intensity using a 4-point scale (0=no headache, 1=mild headache, 2=moderate headache, 3=severe headache).

Secondary objectives included evaluating additional efficacy and safety outcomes of Canvert-M in managing migraine attacks.

DETAILED DESCRIPTION:
In this study, participants are asked to:

* Apply an adequate amount of Canvert-M roll-on to the areas of the forehead, temporal, behind the ears, and base of the neck, at the onset of a migraine attack. (If the participant's headache persists after 30 minutes, a second dose can be used.)
* Record the date when the headache occurred.
* Record the severity of the headache at various time points (before using Canvert-M, and then at 30 minutes, 60 minutes, 120 minutes, 4 hours, and 24 hours after using the Canvert-M roll-on) based on the 4-point scale.
* As much as possible, avoid using any other analgesics for two hours after applying Canvert-M. However, if the headache persists after two hours, the participant may use another medication and should record the name(s) of the drug(s) taken.
* Record a general evaluation of the effectiveness of the investigational product using a simple Likert-type verbal scale.

ELIGIBILITY:
Inclusion criteria:

1. Males and females with age of 18 to 55 years
2. Age of migraine onset ˂ 50 years
3. Having a diagnosis of migraine according to the International Classification of Headache Disorders 3rd edition (ICHD-3) for at least one year
4. Having a history of 2-8 attacks per month
5. Remaining stable on prophylactic medication (if used) during the 2 months prior to screening and throughout the study period
6. Using effective contraception by the women of childbearing potential during the study
7. Ability to provide written, informed consent and to be compliant with the schedule of protocol assessments

Exclusion criteria:

1. Having a diagnosis of other primary (cluster and tension) and secondary headache disorders
2. Having a history of chronic migraine headache
3. History of resistant or refractory migraine headaches based on European Headache Federation consensus
4. Receiving any abortive medication for the treatment of migraine within 48 hours before using Canvert-M
5. History of psychiatric and neurologic disorders (except migraine) or any medical comorbid conditions that interfere with the study results
6. History of nasal sensitivity or allergy to menthol, lavender, rosemary, eucalyptus, wintergreen and basil oil
7. The presence of any skin lesions in the areas where the product is used
8. Treatment with any investigational agent within 30 days prior to screening
9. History of substance use disorders
10. Nursing mothers, pregnant women, and women who plan to become pregnant during the study period
11. Taking carbamazepine, cilostazol, citalopram, clarithromycin, clobazam, colchicine, cyclosporine, digoxin, itraconazole, phenobarbital, phenytoin, rifampin, sirolimus, tacrolimus, tizanidine, and warfarin within 14 days of the study procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-09-16 (Estimated); Study Completion 2025-09-16 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants who report improvement in headache pain by at least one severity level (according to the 4-point scale) at 2 hours after treatment, and before the use of any rescue medication. | Pre-treatment and 2 hours after treatment
  4-point scale: 0=no headache, 1=mild headache, 2=moderate headache, 3=severe headache

SECONDARY OUTCOMES:
The percentage of participants who report improvement in headache pain by at least one severity level according to the 4-point scale at 1 hour and 24 hours after treatment compared to pretreatment pain | Pre-treatment, 1 hour and 24 hours after treatment
  4-point scale: 0=no headache, 1=mild headache, 2=moderate headache, 3=severe headache
The percentage of subjects who need rescue medication 2 hours after treatment | 2 hours after treatment
The global evaluation of treatment efficacy based on a simple Likert-type verbal scale asked from the participants | 24 hours after treatment
  Likert-type verbal scale: Very poor, Poor, No opinion, Good, Very good
Safety assessment by evaluation of adverse events (AEs) | From the screening visit and for up to 30 days
  Adverse events (AEs) were assessed at all visits. All reported events were classified as mild, moderate, or severe. Moreover, seriousness of AEs was assessed according to International Council for Harmonization (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran Province, Tehran, Imam Khomeini Street (RA) - Before Hassan Abad Square, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
Data produced in the present study are available upon reasonable request from the investigators.